CLINICAL TRIAL: NCT06016608
Title: Early Screen, Systematic Evaluation and Risk Warning of Polyvascular Disease Based on Multi-modality Imaging
Brief Title: An Imaging Study of Polyvascular Disease
Status: Recruiting | Type: Observational
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yu Bo, Director, Harbin Medical University
Other Study IDs: ChiCTR2300074638
Record Dates: First submitted 2023-08-22; First posted 2023-08-29 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Polyvascular Disease
MeSH Terms: interventions — Magnetic Resonance Angiography; Computed Tomography Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Polyvascular disease
  Interventions: Diagnostic Test: Magnetic Resonance Angiography, Ocular OCTA, CT Angiography

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Angiography, Ocular OCTA, CT Angiography — Magnetic Resonance Angiography of intracranial artery, carotid artery, renal artery and lower extremity artery, CT angiography of coronary artery or intracranial artery

SUMMARY:
1. Establish a multimodality imaging database for PVD, improve the one-stop screening process for early PVD based on artificial intelligence, build a full-cycle control information platform, and promote the construction and standardization of a multidisciplinary co-morbidity and co-management diagnosis and treatment model.
2. Based on non-invasive, zero-contrast ocular OCTA combined with one-stop CTA imaging of the heart and brain, construct an integrated "eye-heart-brain" early warning model for PVD, and explore a potential non-invasive and convenient early warning system for PVD.
3. Based on the multi-omics, investigate EVs-mediated intercellular communication network, elucidate the roles and regulatory mechanisms of EVs in the development of PVD, search for potential targets for intervention, and construct an artificial intelligence-based "pan-vascular score" risk assessment system based on the combination of multi-modality imaging and multi-omics biomarkers.

ELIGIBILITY:
Inclusion Criteria:

Task 1:

1. Patients with coronary artery disease (≥50% stenosis in any coronary artery on coronary angiography)
2. Age ≥18 years old
3. Proposed OCT-IVUS integrated imaging system
4. able to provide written informed consent prior to the start of any procedures related to the study.

Task 2:

1. patients with coronary artery disease (coronary angiography reveals ≥50% degree of stenosis in any coronary artery) and patients with stroke or TIA (confirmed by a neurologist)
2. Age ≥ 18 years
3. able to provide written informed consent prior to the start of any procedures related to the study.

Exclusion Criteria:

Task 1:

1. severely tortuous/calcified coronary arteries with anticipated difficulty in completing the OCT-IVUS integrated imaging system
2. uncontrolled congestive heart failure or acute left heart failure;plan
3. claustrophobia;
4. left main stem occlusion;
5. proposed coronary artery bypass grafting (CABG);
6. uncontrolled severe ventricular arrhythmia;
7. active bleeding or severe bleeding tendency;
8. acute stroke;
9. patients with hemodynamic instability or unstable cardiac electrical activity (including shock) ;
10. severe renal insufficiency and/or anuria, except in cases where dialysis treatment has been planned;
11. contraindications to the application of contrast media;
12. patients who are severely uncooperative due to psychiatric or serious systemic illness;
13. Patients who, in the opinion of the investigator, are unsuitable for participation in the study.

Task 2:

1. patients who are unable to comply with the follow-up schedule;
2. uncontrolled congestive heart failure or acute left heart failure;
3. patients with a life expectancy of less than 6 months;
4. left main stem occlusion;
5. proposed coronary artery bypass grafting (CABG);
6. uncontrolled severe ventricular arrhythmia;
7. active bleeding or severe bleeding tendency;
8. patients with hemodynamic instability or unstable cardiac electrical activity (including shock) ;
9. severe renal insufficiency and/or anuria, except in cases where dialysis treatment has been planned;
10. contraindications to the application of contrast media;
11. patients who are severely uncooperative due to psychiatric or serious systemic illness;
12. patients who, in the opinion of the investigator, are not suitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with polyvascular disease in the 2nd Affiliated Hospital of Harbin Medical University
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Task1: MACE | 1 year
  All cause death, stroke, myocardial reinfarction, unplanned revascularization, lower extremity artery disease
Task2: Plaque characteristics | 1 year
  Plaque morphology on OCT

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Jia, MD. Ph.D, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No